CLINICAL TRIAL: NCT03115203
Title: Morphometric Study of the Muscles of the Skin in MRI 3 Tesla in Patients With Facial Paralysis.
Acronym: SIMOVI IRM 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0013
Record Dates: First submitted 2017-03-31; First posted 2017-04-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Facial Paralysis
Keywords: muscle skin; IRM 3 tesla
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial paralysis (Other)
  Interventions: Other: Carry out the morphometric evaluation of the muscles of the skin, especially the large zygomatic muscle, in patients with sequelae of facial paralysis
- Healthy subject (Other)
  Interventions: Other: Carry out the morphometric evaluation of the muscles of the skin, especially the large zygomatic muscle, in healthy subjects

INTERVENTIONS:
Other: Carry out the morphometric evaluation of the muscles of the skin, especially the large zygomatic muscle, in patients with sequelae of facial paralysis — Carry out the morphometric evaluation of the muscles of the skin, especially the large zygomatic muscle, in patients with sequelae of facial paralysis
  Arms: Facial paralysis
Other: Carry out the morphometric evaluation of the muscles of the skin, especially the large zygomatic muscle, in healthy subjects — Carry out the morphometric evaluation of the muscles of the skin, especially the large zygomatic muscle in healthy subjects (data obtained from the SIMOVI project being published).
  Arms: Healthy subject

SUMMARY:
The problem posed is the possibility of objectively assessing facial muscle mobility.

Today, in patients with facial paralysis, the assessment of the deficit is carried out using a subjective scale such as the House Brackman [1] or EMG scale of the facial nerve but does not distinguish each muscle individually . Objective measurements of skin muscles such as thickness and volume, in preoperative assessment of a facial paralysis rehabilitation surgery, would be useful in order to choose the most appropriate surgical technique. Indeed, too much amyotrophy will contraindicate hypoglosso-facial anastomosis (VII-XII) and it will be preferable to propose a temporal elongation myoplasty or a reinfused free muscle flap.

Similarly, it would be useful to be able to objectively evaluate the recovery of muscle function after facial allo-transplantation.

Although electromyography has been developed since the work of Duchenne de Boulogne, little research has been carried out on the development of noninvasive methods to objectively characterize in vivo skin muscles (variation, position, orientation, morphometry). The main morphometric data of the skin muscles come from anatomical dissections.

Imaging of the skin muscles has not been specifically developed. Some studies have been carried out to visualize these muscles in MRI 1.5 Tesla in pathologies such as myasthenia gravis, facial paralysis, and labio-alveolo-palatine clefts for example.

The originality of the project is to develop a method allowing to establish a quantitative correlation between the movements of the face and the muscular changes. This correlation will be achieved by associating muscular morphological data derived from MRI acquisitions and cutaneous deformations resulting from clinical examinations. This non-invasive approach should make it possible to establish objective and reproducible indicators in patients with facial paralysis sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Subject, for which a diagnosis of facial paralysis has been made, female or male, over 18 years of age.

Exclusion Criteria:

* Pregnancy and lactation,
* a patient with a contra-indication to MRI (Claustrophobia, Pace Maker, Neurosurgical Clips, Vascular Clips, Cardiac Valves, V.peritoneal Valves, Cochlear Implant, Neuro-Stimulator, Intra-Orbital Metal Shards (Articular Prosthesis, Dental Prosthesis, Contact Glass, Insulin Pumps, Intrauterine Device, Tattoo, Piercing / Implants.))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2023-08-08 (Estimated); Study Completion 2023-08-08 (Estimated)

PRIMARY OUTCOMES:
The measurement of the volume of the large zygomatic muscle in patients with facial paralysis compared to the mean volume of the large zygomatic muscle in healthy subjects. | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France